CLINICAL TRIAL: NCT07239193
Title: Effect of Demineralized Dentin Matrix Versus Mineralized Plasmatic Matrix on Alveolar Ridge Preservation in Molar Extraction Sites; A Randomized Clinical Trial.
Brief Title: Demineralized Dentin Matrix Versus Mineralized Plasmatic Matrix on Alveolar Ridge Preservation in Molar Extraction Sites
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Suliman Ahmed Badr, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DDM in socket preservation
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Socket Preservation; Alveolar Ridge Preservation
Keywords: socket preservation; alveolar ridge preservation; DDM; demineralized dentin matrix; MPM; mineralized plasmatic matrix
MeSH Terms: interventions — Demineralized Dentin Matrix; DDMS

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups in a 1:1 ratio.
  Group A will receive socket grafting with autogenous Demineralized Dentin Matrix (DDM) mixed with Platelet-Rich Fibrin (PRF), while Group B will receive Mineralized Plasmatic Matrix (MPM) composed of xenograft mixed with Platelet-Rich Plasma (PRP). Each participant will receive only one type of intervention.
Who Masked: Participant, Outcomes Assessor
Masking Description: Single-blind design - participants will not be informed which grafting material (DDM or MPM) was used in their treatment. The operating surgeons and data analysts will be aware of the allocation due to the nature of the procedures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Demineralized Dentin Matrix (DDM) + Platelet-Rich Fibrin (PRF) (Experimental): Participants in this group will receive socket grafting using Demineralized Dentin Matrix (DDM) prepared from their own extracted tooth. The dentin is cleaned, ground into particles, demineralized using 0.6 N hydrochloric acid, rinsed with saline, and mixed with autologous Platelet-Rich Fibrin (PRF) before being placed into the extraction socket. The socket is then closed with resorbable sutures for healing.
  Interventions: Biological: Demineralized Dentin Matrix (DDM) + Platelet-Rich Fibrin (PRF)
- Mineralized Plasmatic Matrix (MPM) (Active Comparator): Participants in this group will receive socket grafting using a Mineralized Plasmatic Matrix (MPM) composed of a commercially available xenograft mixed with Platelet-Rich Plasma (PRP). The mixture forms a cohesive mineralized matrix that is placed into the extraction socket and stabilized with sutures.
  Interventions: Biological: Mineralized Plasmatic Matrix (MPM)

INTERVENTIONS:
Biological: Demineralized Dentin Matrix (DDM) + Platelet-Rich Fibrin (PRF) — Autogenous dentin-derived grafting material is used as a bone substitute for alveolar ridge preservation following molar extraction. PRF, obtained from the patient's centrifuged blood, is mixed with DDM to enhance graft stability and promote healing.
  Arms: Demineralized Dentin Matrix (DDM) + Platelet-Rich Fibrin (PRF)
Biological: Mineralized Plasmatic Matrix (MPM) — A xenogenic bone substitute is mixed with autologous platelet-rich plasma to form a mineralized plasmatic matrix, which serves as a control graft for ridge preservation after molar extraction.
  Arms: Mineralized Plasmatic Matrix (MPM)

SUMMARY:
When a tooth is removed, the bone around it (called the alveolar ridge) naturally shrinks. This study compares two bone grafting materials to find out which one better preserves bone after molar extraction:

Demineralized Dentin Matrix (DDM): A material made from the patient's own extracted tooth, treated to remove minerals while keeping bone-forming proteins.

Mineralized Plasmatic Matrix (MPM): A mixture of a standard bone substitute and platelet-rich plasma from the patient's blood.

DETAILED DESCRIPTION:
Alveolar ridge resorption is a predictable biological process following tooth extraction, particularly in molar sites where the bone structure is more complex. Maintaining ridge volume is essential for optimal future implant placement and prosthetic rehabilitation. Various grafting materials and biologic enhancers have been used to minimize post-extraction bone loss; however, cost, availability, and biocompatibility remain significant challenges, especially with xenograft and allograft materials.

This randomized clinical trial investigates and compares two autogenous and biologically enhanced approaches for alveolar ridge preservation following molar extraction. The first method utilizes Demineralized Dentin Matrix (DDM) prepared from the patient's own extracted tooth. DDM provides a naturally derived scaffold rich in collagen and bone morphogenetic proteins (BMPs), offering both osteoconductive and osteoinductive potential. The second method uses a Mineralized Plasmatic Matrix (MPM), a combination of a xenograft bone substitute mixed with Platelet-Rich Plasma (PRP), which represents a widely used regenerative option in oral surgery.

The study is designed as a parallel-group, single-blind, randomized clinical trial conducted at the Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Cairo University. Eligible adult patients requiring extraction of non-restorable multi-rooted molars will be enrolled and allocated equally into two groups. Both groups will undergo atraumatic extraction followed by immediate socket grafting with either DDM+PRF or MPM+PRP.

Standardized postoperative care will be provided to all participants, and healing will be monitored both clinically and radiographically. Cone-beam computed tomography (CBCT) will be used to evaluate alveolar bone width, height, and density immediately after extraction and at 4 months postoperatively. Pain and soft-tissue healing will also be assessed using validated clinical indices.

The study's primary objective is to determine whether Demineralized Dentin Matrix (DDM) provides superior preservation of alveolar ridge dimensions and bone quality compared to Mineralized Plasmatic Matrix (MPM) in molar extraction sites. The hypothesis tested is that there will be no significant difference between both materials regarding bone preservation and regeneration outcomes.

This trial is expected to provide evidence supporting the clinical viability of using recycled autogenous tooth material as a cost-effective and biocompatible alternative to commercially available xenografts, potentially expanding regenerative options for clinicians and improving access to affordable biologic grafting solutions.

ELIGIBILITY:
Inclusion Criteria:

- Non-restorable tooth indicated for extraction Multi-rooted teeth Age group of 18 to 55 years Patients free from any systemic disease that may affect bone healing.

Exclusion Criteria:

- Pregnant females Active infection at extraction site Smokers Systemic conditions affecting healing (e.g. diabetes, medications as bisphosphonates...) Poor oral hygiene. Patient with systemic disease that may affect bone healing. o Uncooperative patient.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Alveolar Ridge Width | Baseline (immediately postoperative) and 4 months postoperatively.
  Measurement of horizontal bone width at the extraction site using cone-beam computed tomography (CBCT).

SECONDARY OUTCOMES:
Change in Alveolar Ridge Height | Baseline (immediately postoperative) and 4 months postoperatively.
  Measurement of vertical bone height at the extraction site using CBCT.
Change in Bone Density | Baseline (immediately postoperative) and 4 months postoperatively.
  Evaluation of bone density in the grafted socket area using CBCT grayscale values.
Postoperative Pain | 2 days, 1 week, and 1 month postoperatively.
  Subjective evaluation of pain intensity at the surgical site using the Visual Analogue Scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Ibrahim ElGhareeb, Phd, Study Chair — Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, Cairo University; Salah Eldin ElAbbasy, Phd, Study Director — Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, Cairo University; Ahmed Suliman Ahmed, Bds, Principal Investigator — Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University - Department of Oral and Maxillofacial Surgery, Cairo, Egypt